CLINICAL TRIAL: NCT00028002
Title: A Phase II Trial of Neoadjuvant/Adjuvant STI-571 (Gleevec NSC #716051) for Primary and Recurrent Operable Malignant GIST Expressing the KIT Receptor Tyrosine Kinase (CD117)
Brief Title: Neoadjuvant and Adjuvant Imatinib Mesylate in Treating Patients With Primary or Recurrent Malignant Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: American College of Radiology Imaging Network (Network); Eastern Cooperative Oncology Group (Network); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02437; NCI-2012-02437 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-RTOG-R0132; RTOG S-0132; ACRIN-6665 (Other: CIP); CDR0000069111 (CIP); RTOG-S-0132; RTOG-0132 (Other: Radiation Therapy Oncology Group); RTOG-0132 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (1):
- Arm I (Experimental): Patients receive oral imatinib mesylate once daily. Treatment continues for 8 weeks in the absence of disease progression. Patients with disease progression are considered for immediate surgical resection. Otherwise, after 8 weeks, patients undergo surgical resection to debulk all gross tumor. Two to four weeks after surgery, patients receive oral imatinib mesylate once daily for 2 years.
  Interventions: Procedure: Conventional Surgery; Drug: Imatinib Mesylate

INTERVENTIONS:
Procedure: Conventional Surgery — Undergo surgical resection
Drug: Imatinib Mesylate — Given orally
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571

SUMMARY:
Phase II trial to study the effectiveness of neoadjuvant and adjuvant imatinib mesylate in treating patients who are undergoing surgery for primary or recurrent malignant gastrointestinal stromal tumor. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving imatinib mesylate before and after surgery may shrink the tumor so it can be removed and may kill any tumor cells remaining after surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the progression-free survival of patients with primary or recurrent potentially resectable malignant gastrointestinal stromal tumor treated with neoadjuvant and adjuvant imatinib mesylate.

II. Determine the objective response rate of patients treated with this drug. III. Determine the safety of this drug in these patients.

OUTLINE:

Patients receive oral imatinib mesylate once daily. Treatment continues for 8 weeks in the absence of disease progression. Patients with disease progression are considered for immediate surgical resection. Otherwise, after 8 weeks, patients undergo surgical resection to debulk all gross tumor. Two to four weeks after surgery, patients receive oral imatinib mesylate once daily for 2 years.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant gastrointestinal stromal tumor

  * Potentially resectable primary disease
  * Potentially resectable recurrent disease

    * Local or intra-abdominal/pelvic metastatic disease
* Documented c-kit (CD117) expression by immunohistochemical analysis of either initial core specimen or, if recurrent disease, from original tumor block
* Primary disease must be visceral, intra-abdominal, or pelvic in origin
* At least 1 unidimensionally measurable lesion

  * At least 5 cm for primary disease
  * At least 2 cm for recurrent disease
* At least 1 viable core biopsy tumor specimen obtained within 8 weeks before registration
* Performance status - Zubrod 0-2
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT/AST no greater than 2.5 times ULN
* No uncontrolled chronic liver disease
* Creatinine no greater than 1.5 times ULN
* No uncontrolled chronic renal disease
* No New York Heart Association class III or IV cardiac disease
* Must be able to lie still in the PET scanner for approximately 1-2 hours
* No uncontrollable hyperglycemia
* No medical or psychological condition that would preclude study participation
* No severe or uncontrolled medical disease
* No active uncontrolled infection
* No known or suspected hypersensitivity to any component of the study drug
* Any prior malignancy is allowed provided patient remains disease free from that malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* At least 28 days since prior biologic therapy
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* At least 28 days since prior chemotherapy
* At least 28 days since prior radiotherapy
* See Disease Characteristics
* At least 28 days since prior investigational drugs
* At least 28 days since prior imatinib mesylate
* No concurrent therapeutic doses of warfarin
* Concurrent low-molecular weight heparin or mini-dose warfarin (1 mg per day) prophylaxis is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2002-03-31 (Actual); Primary Completion 2009-01-28 (Actual); Study Completion 2009-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burton Eisenberg, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Radiation Therapy Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Van den Abbeele AD, Gatsonis C, de Vries DJ, Melenevsky Y, Szot-Barnes A, Yap JT, Godwin AK, Rink L, Huang M, Blevins M, Sicks J, Eisenberg B, Siegel BA. ACRIN 6665/RTOG 0132 phase II trial of neoadjuvant imatinib mesylate for operable malignant gastrointestinal stromal tumor: monitoring with 18F-FDG PET and correlation with genotype and GLUT4 expression. J Nucl Med. 2012 Apr;53(4):567-74. doi: 10.2967/jnumed.111.094425. Epub 2012 Mar 1. PMID 22381410
- [Result] Eisenberg BL, Harris J, Blanke CD, Demetri GD, Heinrich MC, Watson JC, Hoffman JP, Okuno S, Kane JM, von Mehren M. Phase II trial of neoadjuvant/adjuvant imatinib mesylate (IM) for advanced primary and metastatic/recurrent operable gastrointestinal stromal tumor (GIST): early results of RTOG 0132/ACRIN 6665. J Surg Oncol. 2009 Jan 1;99(1):42-7. doi: 10.1002/jso.21160. PMID 18942073
- [Result] Wang D, Zhang Q, Blanke CD, Demetri GD, Heinrich MC, Watson JC, Hoffman JP, Okuno S, Kane JM, von Mehren M, Eisenberg BL. Phase II trial of neoadjuvant/adjuvant imatinib mesylate for advanced primary and metastatic/recurrent operable gastrointestinal stromal tumors: long-term follow-up results of Radiation Therapy Oncology Group 0132. Ann Surg Oncol. 2012 Apr;19(4):1074-80. doi: 10.1245/s10434-011-2190-5. Epub 2011 Dec 28. PMID 22203182

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib Mesylate: Patients receive oral imatinib mesylate once daily. Treatment continues for 8 weeks in the absence of disease progression. Patients with disease progression are considered for immediate surgical resection. Otherwise, after 8 weeks, patients undergo surgical resection to debulk all gross tumor. Two to four weeks after surgery, patients receive oral imatinib mesylate once daily for 2 years.
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 63
Completed | 52 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 11
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible | 8

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 58.5 [24.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Rate of Disease Progression at 2 Years
Description: Kaplan-Meier estimate of disease progression rate. Disease progression is determined by Response Evaluation Criteria in Solid Tumours criteria (RECIST). RECIST criteria is described here: http://ctep.cancer.gov/protocolDevelopment/docs/recist_guideline.pdf
Time Frame: From registration to two years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 52
percentage of participants | 13.8 [4.2 to 23.4]

2. Secondary Outcome: Rates of Objective Response (Complete, Partial, and Stable)
Description: The percentage of patients who achieved a complete, partial or stable response prior to surgery as assessed by Response Evaluation Criteria in Solid Tumours criteria (RECIST). RECIST criteria is described here: http://ctep.cancer.gov/protocolDevelopment/docs/recist_guideline.pdf.
Time Frame: Pretreatment and prior to surgery (at 4-10 weeks, based on surgery timing)
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 52
percentage of participants
  Complete Response | 0 [0 to 0]
  Partial Response | 5.8 [1.2 to 15.9]
  Stable Disease | 86.5 [74.2 to 94.4]

3. Secondary Outcome: Percentage of Patients With Major Toxicity (Toxicity Grade ≥ 3)
Description: Highest grade toxicity per subject was counted. Toxicities were graded using Common Toxicity Criteria (CTC) v 2.0. Grade refers to the severity of the toxicity, using Grades 1 through 5 with unique clinical descriptions of severity for a given toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity.
Time Frame: Analysis occurs after all patients have been on study for at least 2 years. Measured from start of treatment to end of follow-up, to a maximum of 4.95 years.
Population: All eligible patients who started study treatment (for pre-surgery), and who additionally had surgery (post-surgery)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 52
percentage of participants
  Pre-surgery | 34.6 [22.0 to 49.1]
  Post-surgery: number analyzed (Participants) | 45
  Post-surgery | 48.9 [33.7 to 64.2]

4. Secondary Outcome: FDG-PET as Biological Marker of Metabolic Response(MR) During Imatinib Mesylate (IM) Treatment, in Patients With GIST Who Are naı¨ve to Tyrosine Kinase Inhibitor Therapy
Description: evaluate FDG-PET as a non-invasive functional imaging tool to assess in situ tumor metabolism (as measured by the Standardized Uptake Values of FDG in the tumor) prior to and during the administration of IM. %change in SUVmax <1 indicate decreased tumor metabolism while values >1 indicated an increase in tumor metabolism.
  Metabolic response by 18F-FDG PET was determined in accordance with the criteria of the European Organization for Research and Treatment of Cancer EORTC), with increases or decreases of more than 25% in SUVmax defining progressive metabolic disease (PMD) and partial metabolic response (PMR), respectively, and new lesions defining PMD.
Time Frame: change from baseline to 1 week post therapy
Measure: Mean (Full Range); unit: percentage change in SUVmax
Groups:
- PET Patricipants: FDG-PET was done at baseline, 1-7 days after IM initiation, in patients with GIST undergoing neoadjuvant IM therapy.
  Tumor GLUT4 expression by immunohistochemistry (IHC) and mutation analyses were done at baseline and/or surgery. Background-subtracted SUVmax was measured in all lesions and summed; Metabolic Response (MR)based on EORTC criteria was compared to Response Evaluation Criteria in Solid Tumors (RECIST), GLUT4 expression, and KIT/PDGFRA mutation status.
Arm/Group | PET Patricipants
Number analyzed (Participants) | 44
percentage change in SUVmax | -59.4 [-100 to 81.4]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) information is collected Weeks 1, 4, 8, Months 3,8,9, then every 3 months until 2 years, then every 6 months until 5 years, then annually. (SAE = Serious Adverse Event).
Description: Per the protocol, toxicity data was collected via CTC 2.0 then mapped to CTCAE 4.0 to report here. Subjects experiencing more than one of a given adverse event (AE) are counted only once for that AE.
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 22/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=52)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Cardiac disorders - Other (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Esophageal fistula (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 1
Infections and infestations - Other (Infections and infestations) | 5
Wound infection (Infections and infestations) | 3
Neutrophil count decreased (Investigations) | 4
Serum amylase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
"Respiratory, thoracic and mediastinal disorders - Other" (Respiratory, thoracic and mediastinal disorders) | 1
Capillary leak syndrome (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 3
Vascular disorders - Other (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=52)
Anemia (Blood and lymphatic system disorders) | 44
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 4
Dry eye (Eye disorders) | 3
Eye disorders - Other (Eye disorders) | 2
Watering eyes (Eye disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 10
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 29
Dyspepsia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 5
Gastric ulcer (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 34
Rectal hemorrhage (Gastrointestinal disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 17
Chills (General disorders) | 3
Fatigue (General disorders) | 20
Fever (General disorders) | 7
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 12
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1
Immune system disorders - Other (Immune system disorders) | 1
Infections and infestations - Other (Infections and infestations) | 8
Wound infection (Infections and infestations) | 2
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 17
Blood bilirubin increased (Investigations) | 9
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 6
Investigations - Other (Investigations) | 5
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 21
Platelet count decreased (Investigations) | 15
Serum amylase increased (Investigations) | 1
Weight gain (Investigations) | 6
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 26
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 15
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 5
Vasovagal reaction (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Renal and urinary disorders - Other (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Capillary leak syndrome (Vascular disorders) | 28
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 3
Hypertension (Vascular disorders) | 4
Lymphedema (Vascular disorders) | 3
Vascular disorders - Other (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less